CLINICAL TRIAL: NCT05323643
Title: Role of Ultrasound in Evaluation of Tendon and Ligament Abnormalities in Hand and Fingers
Brief Title: Role of US in Evaluation of Tendon and Ligament Abnormalities in Hand and Fingers
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Wafaa Ahmed Sayed Mohamed Sebaie, Radiology resident at Assiut University Hospitals, Assiut University
Other Study IDs: US in hand & fingers
Record Dates: First submitted 2022-04-05; First posted 2022-04-12 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Tendon Disorder
MeSH Terms: conditions — Tendinopathy | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional

INTERVENTIONS:
Device: Ultrasound — musculoskeletal US will be performed using commercially -available equipment, with high frequency linear -array transducers and a standard gel interface. The higher frequency transducers provide better spatial resolution, while the lower frequency transducers provide a greater depth of tissue penetrance. Colour Doppler US is also performed in most cases as it plays an important role in supporting and confirming diagnoses, by providing valuable information about the pathophysiology of the abnormality.
  The patients will be seated with hands placed on a table, to permit examination of both volar and dorsal aspects, in longitudinal and transversal axis. Examination of the hands and fingers usually requires a large amount of transmission gel, in order to avoid compression and to permit dynamic evaluation. When acute trauma with skin lesions is investigated, sterile transmission gel, or sterile acoustic standoff pads can be used

SUMMARY:
Assessment of the role of USG in the evaluation of tendon and ligament abnormalities in hand and fingers in traumatic & non-traumatic causes.

DETAILED DESCRIPTION:
The hand and fingers are the most important functional parts of the body in daily life activities and are prone to traumatic injuries and susceptible to a wide array of inflammatory diseases. Tendon abnormalities of the hand and the fingers are common disorders, particularly among athletes and in the elderly. These abnormalities may be symptomatic degenerative changes, inflammatory, or rupture. Tendon disorders are a common cause of pain and loss of function. Chronic tendon disorders are much more common than acute injuries and are the result of overuse or age-related tendon degeneration.

There is a wide spectrum of hand and finger pathological conditions that can be demonstrated using Ultrasonography. Superficial structures of the wrist, hand, and fingers, including the tendons, ligaments, nerves, and vessels, are amenable to imaging with high-frequency US. US can depict masses and fluid collections, help locate radiolucent foreign bodies, characterize traumatic or overuse tendon or ligament pathology, and help evaluate compressive peripheral neuropathy and microvascular blood flow. Additionally, this modality improves the accuracy of therapeutic intra-articular or peritendinous injections and facilitates aspiration of fluid collections, such as ganglia.

Due to the improvement of imaging techniques in the last years, the performance of ultrasonography (US) in detecting pathological changes in the musculoskeletal system dramatically increased. Moreover, dynamic examination allows better evaluation of the type and extension of the lesions. An anatomical course of the nerves and tendons can be depicted by US, thus offering valuable information on the exact location and type of possible lesions.

The role of USG in the assessment of tendon disorders is steadily increasing due to its being low cost, fast, wide-spread availability, and non-invasive. Additionally, it may offer a dynamic assessment of the flexor and extensor tendons, collateral ligaments, and supporting structures of the fingers, such as the extensor hood and the volar plate, as well as space-occupying lesions.

The quality of USG assessment of anatomical structures in the hand has highly improved over the last time. The development of high resolution with the highest possible frequency of modern ultrasound equipment and the superficial location of most tendons allows the spectrum of tendon abnormalities to be easily depicted with USG. US facilitates dynamic, real-time evaluation of bones, joints, tendons, nerves, and vessels, making it an ideal imaging modality for hand and finger conditions.

ELIGIBILITY:
Inclusion Criteria:

* Patients complaining of pain or masses of the hands and the fingers or referred for assessment of tendon & ligaments which are involved in such pain and swellings.

Exclusion Criteria:

* Patients with a recent history of local operative intervention will be excluded

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients complaining of pain or masses in hands or fingers, patients with inflammatory conditions, and traumatic injuries.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2023-11-11 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Evaluating the tendon and ligament abnormalities by the US and correlating them with the symptoms. | Baseline
  characterization of tendon and ligament pathologies in hand and fingers in traumatic and non-traumatic causes by using clinical history and imaging appearance by US, one can determine the diagnosis

SECONDARY OUTCOMES:
Assessment of the role of USG in the evaluation of tendon and ligament abnormalities in hand and fingers. | Baseline
  help in the diagnosis of different hand and finger diseases, view of reliability and sensitivity: specificity ratio in assessing tendon and ligament diseases in hand and fingers either in inflammatory conditions or traumatic injuries